CLINICAL TRIAL: NCT05278039
Title: Training Swallowing Initiation During Expiration: Impact on Safety and Efficiency Following Treatment for Oropharyngeal Head and Neck Cancer
Brief Title: Training Swallowing Initiation During Expiration
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Northwestern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Bonnie Martin-Harris, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01CA262502 (NIH)
Record Dates: First submitted 2022-02-08; First posted 2022-03-14 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Head and Neck Cancer; Dysphagia; Oropharyngeal Dysphagia; Oropharynx Squamous Cell Carcinoma
Keywords: Dysphagia; Swallowing Disorders; Swallowing Rehabilitation; Telehealth; Wearable Sensor; Respiratory-Swallow Coordination; Modified Barium Swallow Study
MeSH Terms: conditions — Head and Neck Neoplasms; Deglutition Disorders; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Intervention Model Description: Randomized-controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors will be naive to experimental condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Respiratory-Swallow Phase Training (Experimental): Participants will be trained to initiate swallowing during expiration.
  Interventions: Behavioral: Respiratory-Swallow Phase Training
- Swallow Practice (Sham Comparator): Participants will practice swallowing, but will not learn the key therapeutic element (i.e., initiating swallowing during expiration).
  Interventions: Other: Swallow Practice

INTERVENTIONS:
Behavioral: Respiratory-Swallow Phase Training — Participants will complete 6 respiratory-swallow phase training sessions that will last approximately one hour.
  Arms: Respiratory-Swallow Phase Training
Other: Swallow Practice — Participants will complete 6 "swallow practice" sessions that will last approximately one hour.
  Arms: Swallow Practice

SUMMARY:
Head and neck cancers have escalated to epidemic levels in the United States, and survivors are suffering from life-long, devastating swallowing disorders with limited therapeutic options. This clinical trial investigates a novel swallowing treatment that trains initiation of swallowing during the expiratory phase of respiration to improve swallowing safety and efficiency.

DETAILED DESCRIPTION:
Head and neck cancers (HNC) have increased to epidemic levels in the United States. Despite good response to cancer treatment, survivors are suffering life-long toxicities that result in swallowing problems (dysphagia). Treatment options for dysphagia after HNC are extremely limited, focus on swallowing movements alone, and do not consider the importance of respiratory-swallow phase patterning. Prior evidence has demonstrated that when aberrant respiratory-swallow phase patterning is present (initiation of swallowing during inspiration) in patients with HNC, there is a higher occurrence of swallowing impairments, increased residue, and airway invasion. Further, it has been well established that the expiratory limb of the respiratory cycle provides a biomechanically advantageous set point in which to initiate safe and efficient swallowing. This randomized, controlled, Phase II clinical trial examines if respiratory-swallow phase training improves airway protection and swallowing efficiency in HNC survivors who are three or more months post-completion of first-line cancer treatment. The primary goal (Aim 1) is to determine if respiratory-swallow phase training results in increased frequency (%) of swallows initiated during expiration and improved swallowing safety. The secondary goal (Aim 2) is to examine the impact of respiratory-swallow phase training on the frequency of swallows initiated during expiration in wakeful, naturalistic swallowing environments, including eating and drinking. The investigators will recruit 88 HNC survivors with dysphagia, impaired respiratory-swallow phase patterning, and airway compromise. The investigators will deliver therapy remotely using a telehealth platform and an innovative wearable sensor that provides real-time visual feedback of respiratory-swallow movements. Endpoints will be measured from synchronized videofluoroscopic and respiratory-swallow sensor recordings at baseline, within 1-week post-treatment, and 1-month and 3-months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary head and neck cancer
* Three or more months post-completion of first-line cancer treatment
* English speaking
* Functional/corrected visual and hearing acuity
* No current alcohol or other drug abuse
* Without very severe (forced expiratory volume; FEV) 1 <30% predicted) stage Chronic Obstructive Pulmonary Disease (COPD) based on Pulmonary Function Testing (PFT)
* No skin allergy to the medical-grade sensor adhesive
* Tolerate wearing the sensor for at least 10 hours/day
* Tolerate some liquid oral intake on a routine basis
* Normal dexterity to self-administer liquids via teaspoon
* Initiation of swallowing during inspiratory phase of respiration on ≥20% of swallows
* Penetration Aspiration Scale (PAS) score ≥3 or impairment on at least one MBSImP OI score (laryngeal vestibular closure ≥1, tongue base retraction ≥2, or pharyngeal residue ≥2) on at least one swallow during lateral view of MBSS
* A PAS score of ≤6 on at least one liquid consistency without the use of a compensatory strategy or swallow maneuver

Exclusion Criteria:

* Persistent or recurrent cancer at the time of enrollment
* Known allergy to contrast materials or liquids used during the MBSS or training
* Known allergy to sensor adhesive
* Unable to demonstrate competency with the user-friendly technology
* Diagnosis of neurological disorders
* Indwelling tracheostomy tube
* Nasogastric (NG) feeding tube
* History of aspiration pneumonia within the past 12 months
* Unable to self-administer liquid boluses
* Unable to swallow some liquids without a maneuver
* Likely or currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-05-19 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in frequency (%) of swallows initiated during expiration | Change from baseline to 1-week post-treatment and 2-4-6-8-10-12-weeks post-treatment.
  Determines percent (frequency) of the target (expiratory phase) for each swallow.
Change in Penetration-Aspiration Scale scores | Change from baseline to 1-week post-treatment, 1-month post-treatment, and 3-months post treatment. Scores range from 1-8 and higher scores indicate worse outcome.
  Measures presence, depth and reaction to penetration and aspiration.

SECONDARY OUTCOMES:
Change in Normalized Residue Ratio Scale scores | Change from baseline to 1-week post-treatment, 1-month post-treatment, and 3-months post treatment. Scores range from 0 to 100% and higher scores indicate worse outcome.
  Quantifies pharyngeal space residue obtained in the lateral view during Modified Barium Swallow Study (MBSS)
Change in Modified Barium Swallow Impairment Profile (MBSImP) scores | Change from baseline to 1-week post-treatment, 1-month post-treatment, and 3-months post treatment. Oral Total scores range from 0-22 and Pharyngeal Total scores range from 0-26 and higher values indicate worse outcome.
  Measures physiologic swallowing impairment from observations of MBSS recordings

OTHER OUTCOMES:
Change in M.D. Anderson Dysphagia Inventory (MDADI) scores | Change from baseline to 1-week post-treatment, 1-month post-treatment, and 3-months post treatment. Scores range from 20 to 100 and higher scores indicate worse outcome.
  Evaluates the impact of dysphagia on the quality of life of patients with head and neck cancer

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Martin-Harris, PhD, Principal Investigator — Northwestern Memorial Hospital
Locations (2):
- United States (2):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Northwestern University, Evanston, Illinois

IPD SHARING:
Plan to Share IPD: No